CLINICAL TRIAL: NCT04810234
Title: Functional Neural Correlates of Transcutaneous Vagal Nerve Stimulation: Effects of Anatomical Site and Waveform Parameters - An Exploratory High Resolution fMRI Study in Healthy Volunteers
Brief Title: Neural Correlates of tVNS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wingate Institute of Neurogastroenterology (Other)
Responsible Party: Sponsor
Other Study IDs: 65751.068.2018; METC183019 (Other: METC aZM/UM)
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: fMRI; Transcutaneous Vagal Nerve Stimulation (tVNS); Nucleus of the Solitary Tract (NTS)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transcutaneous vagal nerve stimulation (tVNS) — Cervical and auricular transcutaneous stimulation of the vagus nerve

SUMMARY:
Transcutaneous vagal nerve stimulation (tVNS) has been applied to a number of disease areas including visceral pain, depression, cluster headache and Alzheimer's disease. However, there is marked heterogeneity in these studies pertaining to i) the anatomical site of stimulation (neck, inner concha or tragus of ear), and ii) the waveform parameters of the stimulating impulse. This exploratory cross-sectional study will address these knowledge gaps by comparative functional neuroimaging of the neural correlates of tVNS with disparate anatomical sites and electrical waveform characteristics during rest in healthy participants.

ELIGIBILITY:
Inclusion criteria:

* Of female sex;
* Healthy participants (defined as those without a pre-existing medical comorbidity)
* Age between 18 and 40 years;
* BMI between 18 and 30 kg/m2;
* Women on oral contraceptives only
* All subjects should be right-handed.
* Inclusion will be determined on the basis of availability. Subjects should be able to attend for 2 scanning sessions.

Exclusion criteria

* Presence of metallic prostheses, pacemakers, metal clips on blood vessels, metal parts in the eye, an intrauterine device, metal braces, tattoos and/or other metal objects;
* History of major head trauma or head/brain surgery;
* History of claustrophobia;
* History of severe or chronic cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, haematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol;
* Use of regular medication, including vitamin and iron supplementation, except oral contraceptives, within 14 days prior to start of the study;
* Pregnancy, lactation, wish to become pregnant;
* High alcohol consumption (>15 alcoholic units consumed per week);
* Using drugs of abuse;
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study;
* Participants unable to provide informed consent
* Participants with any systemic disease or medications that may influence the autonomic nervous system (e.g. beta-agonists or Parkinson's disease)
* Current smokers or current use of nicotine in any other way (including E-cigarettes and patches)
* History of clinical anxiety or depression, or a hospital anxiety or depression score >8
* Participants whom score 8 or more on the HADS-questionnaire at study commencement
* Patient whom have cardiovascular conduction problems
* Patient with cochlear implants
* Not meeting any of the inclusion criteria above
* Any evidence of structural brain abnormalities examined by anatomical MRI will lead to exclusion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females only (in order to limit confounding)
Study Population: Female healthy volunteers aged between 18-40 years
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) signal activity in the CAN during tVNS | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure

SECONDARY OUTCOMES:
Voxel-wise dependent BOLD signal activity in the NTS of the brainstem; somatosensory cortex; insular cortex; ACC, hypothalamus; thalamus and amygdala during auricular tVNS (parameter set 1) | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure
Voxel-wise dependent BOLD signal activity in the NTS of the brainstem; somatosensory cortex; insular cortex; ACC, hypothalamus; thalamus and amygdala during cervical tVNS )(parameter set 1) | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure
Voxel-wise dependent BOLD signal activity in the NTS of the brainstem; somatosensory cortex; insular cortex; ACC, hypothalamus; thalamus and amygdala during auricular tVNS (parameter set 2) | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure
Voxel-wise dependent BOLD signal activity in the NTS of the brainstem; somatosensory cortex; insular cortex; ACC, hypothalamus; thalamus and amygdala during cervical tVNS (parameter set 2) | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure
Voxel-wise dependent BOLD signal activity in the NTS of the brainstem; somatosensory cortex; insular cortex; ACC, hypothalamus; thalamus and amygdala during subliminal auricular tVNS (parameter set 1) | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure
Functional connectivity / Network Connectivity of CAN regions during "active tVNS" block [to all 5 points as identified above] | During stimulation (difference between stim on - stim off blocks)
  fMRI related outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Maastricht University Medical Center, Maastricht, Netherlands
- Queen Mary University of London. Wingate Institute of Neurogastroenterology, London, United Kingdom